CLINICAL TRIAL: NCT02255474
Title: Soft Bifocal Contact Lens Myopia Control
Brief Title: Bifocal Lenses In Nearsighted Kids
Acronym: BLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Houston (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Jeffrey J. Walline, OD PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014H0231; U10EY023208 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Refractive Errors
Keywords: pediatrics; refractive error - myopia; contact lenses; intervention
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biofinity (Active Comparator): Soft spherical contact lens
  Interventions: Device: Biofinity
- Biofinity Multifocal D +1.50 add (Experimental): The Biofinity Multifocal "D" with a +1.50 add is a soft bifocal contact lens that has a medium reading power
  Interventions: Device: Biofinity Multifocal D +1.50 add
- Biofinity Multifocal D +2.50 add (Experimental): The Biofinity Multifocal "D" with a +2.50 add is a soft bifocal contact lens that has a strong reading power
  Interventions: Device: Biofinity Multifocal D +2.50 add

INTERVENTIONS:
Device: Biofinity Multifocal D +1.50 add — This is a monthly disposable contact lens commercially available from CooperVision
  Arms: Biofinity Multifocal D +1.50 add
Device: Biofinity Multifocal D +2.50 add — This is a monthly disposable contact lens commercially available from CooperVision
  Arms: Biofinity Multifocal D +2.50 add
Device: Biofinity — This is a monthly disposable spherical contact lens commercially available from CooperVision
  Arms: Biofinity

SUMMARY:
This study will evaluate the use of two different bifocal contact lens add powers to prevent further nearsighted progression in children ages 7 to 11 years old. It is theorized that the profile of the bifocal lenses will decrease the amount of change in nearsightedness that the children experience.

DETAILED DESCRIPTION:
The primary goal of this project is to determine whether a commercially available soft bifocal contact lens with a distance-center design can slow myopia progression in children. Using soft bifocal contact lenses to manipulate the peripheral optics of the eye is a novel use for a standard contact lens that may keep children from becoming as nearsighted as they would otherwise. Secondary goals are to determine whether the amount of myopic defocus imposed on the peripheral retina by soft bifocal contact lenses is associated in a dose-dependent manner with slowed myopic progression and to determine whether peripheral myopic blur acts to slow eye growth locally or globally. These important pieces of information will enable investigators to learn about the role of peripheral optics for regulating eye growth, which could ultimately lead to optimization of optical signals to slow myopia progression. Ultimately, the information could be used to design optical devices to prevent the onset of myopia in young children.

Slowing myopia progression or eventually preventing myopia onset could potentially affect approximately 60 million children in the United States alone. While the consequences of myopia are rarely sight-threatening, the quality of life for myopic patients is negatively affected and the health care costs to treat myopia are astronomical (approximately $4.6 billion in 1990). The National Eye Institute recognizes the need to "evaluate the efficacy of potential treatments for delaying the onset or for slowing the progression of myopia, such as lenses that alter peripheral defocus."

Using a common treatment of myopia (contact lenses) to potentially slow myopia progression and to learn about optical signals that regulate eye growth is a very novel approach to solving a problem that affects a large proportion of people in the United States.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 11 years, inclusive, at baseline examination
* -0.75 to -5.00 D, inclusive, spherical component, cycloplegic autorefraction
* ≤1.00 DC, cycloplegic autorefraction
* ≥ 2.00 D difference between the sphere components of the two eyes (anisometropia), cycloplegic autorefraction
* 0.1 logMAR or better best-corrected visual acuity in each eye
* 0.1 logMAR or better visual acuity OU distance and near with a +2.50 D add contact lens
* +2.50 D add lens provides adequate fit with respect to movement and centration

Exclusion Criteria:

* Eye disease or binocular vision problems (e.g., strabismus, amblyopia, oculomotor nerve palsies, corneal disease, etc.)
* Systemic disease that may affect vision, vision development, or contact lens wear (eg, diabetes, Down syndrome, etc.)
* Previous gas permeable, soft bifocal, or orthokeratology contact lens wear or bifocal/PAL spectacle wear (longer than 1 month of wear)
* Previous or current participation in myopia control studies
* Chronic use of medications that may affect immunity, such as oral or ophthalmic corticosteroids for ocular or systemic diseases
* Issues that may interfere with the ability to participate over the next 3 years

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 294 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Walline, OD, PhD, Study Chair — Ohio State University
Locations (2):
- United States (2):
  - Ohio State University College of Optometry, Columbus, Ohio
  - University of Houston College of Optometry, Houston, Texas

REFERENCES:
- [Derived] Chandler MA, Robich ML, Jordan LA, Mutti DO, Berntsen DA, Fenton R, Day E, Walline JJ; BLINK2 Study Group. Accommodation in Children after 4.7 Years of Multifocal Contact Lens Wear in the BLINK Study Randomized Clinical Trial. Optom Vis Sci. 2023 Jul 1;100(7):425-431. doi: 10.1097/OPX.0000000000002040. Epub 2023 Jun 24. PMID 37369096
- [Derived] Gaume Giannoni A, Robich M, Berntsen DA, Jones-Jordan LA, Mutti DO, Myers J, Shaw K, Walker MK, Walline JJ; BLINK Study Group. Ocular and Nonocular Adverse Events during 3 Years of Soft Contact Lens Wear in Children. Optom Vis Sci. 2022 Jun 1;99(6):505-512. doi: 10.1097/OPX.0000000000001902. Epub 2022 Apr 12. PMID 35413027
- [Derived] Walline JJ, Walker MK, Mutti DO, Jones-Jordan LA, Sinnott LT, Giannoni AG, Bickle KM, Schulle KL, Nixon A, Pierce GE, Berntsen DA; BLINK Study Group. Effect of High Add Power, Medium Add Power, or Single-Vision Contact Lenses on Myopia Progression in Children: The BLINK Randomized Clinical Trial. JAMA. 2020 Aug 11;324(6):571-580. doi: 10.1001/jama.2020.10834. PMID 32780139
- [Derived] Schulle KL, Berntsen DA, Sinnott LT, Bickle KM, Gostovic AT, Pierce GE, Jones-Jordan LA, Mutti DO, Walline JJ; Bifocal Lenses in Nearsighted Kids (BLINK) Study Group. Visual Acuity and Over-refraction in Myopic Children Fitted with Soft Multifocal Contact Lenses. Optom Vis Sci. 2018 Apr;95(4):292-298. doi: 10.1097/OPX.0000000000001207. PMID 29561497
- [Derived] Walline JJ, Gaume Giannoni A, Sinnott LT, Chandler MA, Huang J, Mutti DO, Jones-Jordan LA, Berntsen DA; BLINK Study Group. A Randomized Trial of Soft Multifocal Contact Lenses for Myopia Control: Baseline Data and Methods. Optom Vis Sci. 2017 Sep;94(9):856-866. doi: 10.1097/OPX.0000000000001106. PMID 28737608

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Biofinity | Biofinity Multifocal D +1.50 Add | Biofinity Multifocal D +2.50 Add
Started | 98; 98 eyes | 98; 98 eyes | 98; 98 eyes
Completed | 96; 96 eyes | 96; 96 eyes | 95; 95 eyes
Not Completed | 2; 2 eyes | 2; 2 eyes | 3; 3 eyes
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Biofinity: Single vision soft contact lens
- Biofinity +1.50 D Add: Medium add soft bifocal contact lens (+1.50 Diopter add)
- Biofinity +2.50 D Add: High add soft bifocal contact lens (+2.50 Diopter add)
- Total: Total of all reporting groups
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add | Total
Number analyzed (Participants) | 98 | 98 | 98 | 294
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 98 | 98 | 98 | 294
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (1.1) | 10.3 (1.2) | 10.36 (1.2) | 10.3 (1.2)
Age, Customized [Count of Participants; unit: Participants]
  Age: 7 to 9 years | 39 | 39 | 39 | 117
  Age: 10 to 11 years | 59 | 59 | 59 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 49 | 64 | 177
  Male | 34 | 49 | 34 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 26 | 26 | 77
  Not Hispanic or Latino | 72 | 71 | 71 | 214
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 9 | 7 | 9 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 17 | 7 | 5 | 29
  White | 59 | 75 | 66 | 200
  More than one race | 11 | 7 | 13 | 31
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 98 | 98 | 98 | 294
Site [Count of Participants; unit: Participants]
  Columbus, OH | 49 | 48 | 46 | 143
  Houston, TX | 49 | 50 | 52 | 151
Spherical equivalent [Mean (Standard Deviation); unit: Diopters] — Diopters
  Diopters | -2.46 (0.97) | -2.43 (1.11) | -2.28 (0.90) | -2.39 (1.00)
Axial length [Mean (Standard Deviation); unit: mm] — mm
  mm | 24.45 (0.83) | 24.57 (0.85) | 24.43 (0.74) | 24.48 (0.81)
Peripheral axial length [Mean (Standard Deviation); unit: mm]
  20 degree inferior | 24.27 (0.83) | 24.37 (0.85) | 24.24 (0.74) | 24.29 (0.81)
  20 degree nasal | 24.16 (0.85) | 24.31 (0.95) | 24.15 (0.86) | 24.20 (0.88)
  20 degree superior | 24.38 (0.84) | 24.45 (0.85) | 24.36 (0.79) | 24.40 (0.82)
  20 degree temporal | 24.07 (0.85) | 24.20 (0.84) | 24.06 (0.74) | 24.11 (0.81)
  30 degree inferior | 24.03 (0.81) | 24.13 (0.82) | 24.01 (0.72) | 24.06 (0.78)
  30 degree nasal | 24.08 (0.85) | 24.22 (0.87) | 24.07 (0.79) | 24.13 (0.84)
  30 degree superior | 24.20 (0.86) | 24.25 (0.86) | 24.19 (0.80) | 24.21 (0.84)
  30 degree temporal | 23.69 (0.820) | 23.82 (0.80) | 23.69 (0.73) | 23.73 (0.79)
Peripheral defocus [Mean (Standard Deviation); unit: Diopters]
  40 degree nasal | 2.17 (1.17) | 1.07 (1.30) | 0.44 (1.23) | 1.23 (1.42)
  30 degree nasal | 1.06 (0.84) | 0.16 (1.02) | -0.37 (0.95) | 0.28 (1.10)
  20 degree nasal | 0.54 (0.81) | -0.10 (0.77) | -0.37 (0.75) | 0.02 (0.86)
  20 degree temporal | 0.56 (0.75) | -0.27 (0.79) | -0.86 (0.74) | -0.19 (0.96)
  30 degree temporal | 1.29 (1.06) | 0.27 (1.07) | -0.35 (1.21) | 0.40 (1.30)
  40 degree temporal | 1.92 (1.64) | 1.33 (1.71) | 0.87 (1.64) | 1.37 (1.72)

OUTCOME MEASURES:

1. Primary Outcome: Refractive Error Progression
Description: Refractive error, as measured by cycloplegic autorefraction in both eyes, will be measured yearly to assess the difference in progression between the two soft bifocal treatment lenses (+1.50 D add and +2.50 D add) and the control group (soft spherical contact lenses).
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Diopters
Groups:
- Biofinity: Spherical soft contact lens
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add
Number analyzed (Participants) | 97 | 98 | 97
Diopters | -3.46 (1.20) | -3.32 (1.48) | -2.84 (1.22)
Statistical Analysis 1: Comparison: Biofinity vs Biofinity +1.50 D Add vs Biofinity +2.50 D Add; Both eyes used in analysis adjusting for correlation; Test type: Superiority; p < 0.01, Mixed Models Analysis — Adjusted for multiple comparisons, treatment group p-value; Mean Difference (Final Values) = -1.01

2. Secondary Outcome: Ocular Shape Change and Eye Growth
Description: The outcome of interest is the change in ocular shape and measured by the change in peripheral refractive error in the right eye. The change in peripheral refractive error will be compared among the two treatment groups and the control group to determine whether peripheral defocus changes the shape of the eye globally (across the whole eye) or locally (specific to the region of the eye affected by the defocus).
Time Frame: 3 years
Population: Analysis of peripheral eye length changes with treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add
Number analyzed (Participants) | 97 | 98 | 97
mm
  20 degree inferior | 24.92 (0.85) | 24.94 (0.97) | 24.64 (0.79)
  20 degree nasal | 24.86 (0.87) | 24.90 (1.09) | 24.60 (0.93)
  20 degree superior | 24.98 (0.89) | 24.98 (0.97) | 24.74 (0.84)
  20 degree temporal | 24.98 (0.89) | 24.98 (0.97) | 24.71 (0.84)
  30 degree inferior | 24.64 (0.83) | 24.68 (0.94) | 24.45 (0.78)
  30 degree nasal | 24.70 (0.84) | 24.79 (1.01) | 24.51 (0.87)
  30 degree superior | 24.76 (0.92) | 247.77 (0.95) | 24.58 (0.86)
  30 degree temporal | 24.30 (0.82) | 24.29 (0.91) | 24.04 (0.81)
Statistical Analysis 1: Comparison: Biofinity vs Biofinity +1.50 D Add; Individual subject eye length profiles were fit using quadratic equations as a function of gaze angle. The analysis of quadratic coefficients included treatment group, study year (categorical variable), and their interaction adjusted for age, study site, and ethnicity; Test type: Superiority; p = 0.05, Mixed Models Analysis; quadratic coefficient = 0.02

3. Secondary Outcome: Association of Peripheral Defocus to Myopic Progression
Description: Peripheral defocus will be measured in 10 areas (Nasal and temporal zones at 20, 30, and 40 degrees, and superior and inferior zones at 20 and 30 degrees) and analyzed for its relation to myopia progression (as measured by cycloplegic autorefraction in the right eye only).
Time Frame: 3 years
Population: outcome is three-year change in refractive error as a function of baseline peripheral defocus
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add
Number analyzed (Participants) | 97 | 98 | 97
Diopters | -1.01 (0.66) | -0.85 (0.82) | -0.56 (0.66)
Statistical Analysis 1: Comparison: Biofinity vs Biofinity +1.50 D Add vs Biofinity +2.50 D Add; This analysis looks at the three-year change in spherical equivalent refractive error for different eccentricities of peripheral defocus measured with contact lenses in place; Test type: Superiority; p = 0.05, Regression, Linear; Models control for age, sex, axial length at baseline, race, treatment group, treatment group by race interaction; regression coefficient = -0.12

4. Secondary Outcome: Axial Length Progression
Description: Axial length progression, as measured by Lenstar in both eyes, will be measured yearly to assess the difference in progression between the two soft bifocal treatment lenses (+1.50 D add and +2.50 D add) and the control group (soft spherical contact lenses).
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add
Number analyzed (Participants) | 97 | 98 | 97
mm | 25.08 (0.85) | 25.12 (0.97) | 24.81 (0.83)
Statistical Analysis 1: Comparison: Biofinity vs Biofinity +1.50 D Add vs Biofinity +2.50 D Add; Both eyes used in the analysis controlling for the correlation; Test type: Superiority; p = 0.05, Mixed Models Analysis — Adjusted for multiple comparisons; Mean Difference (Final Values) = 0.62

ADVERSE EVENTS:
Time Frame: Three years
Description: Any event, ocular or non-ocular, regardless of relation to contact lens wear that occurred.
Arm/Group | Biofinity | Biofinity +1.50 D Add | Biofinity +2.50 D Add
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 72/97 | 71/98 | 75/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biofinity (N=97) | Biofinity +1.50 D Add (N=98) | Biofinity +2.50 D Add (N=97)
SEAL (Eye disorders) | 3 (3) | 1 (1) | 1 (1) — Superior Epithelial Arcuate Lesion
CLARE (Eye disorders) | 1 (1) | 1 (1) | 2 (2) — Contact lens associated red eye
Corneal epithelial defect (Eye disorders) | 2 (2) | 2 (2) | 5 (5)
Infiltrative keratitis (Eye disorders) | 5 (6) | 4 (5) | 2 (2)
Probable microbial keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Sterile Corneal Ulcer (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Toxic exposure (Eye disorders) | 4 (4) | 3 (3) | 0 (0) — gas. soap in eye
Giant papillary conjunctivitis (Eye disorders) | 3 (3) | 5 (5) | 3 (3)
Ocular allergies (Eye disorders) | 9 (9) | 12 (12) | 22 (25)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Hordeolum/chalazion (Eye disorders) | 9 (10) | 3 (3) | 7 (10)
Eyelash issue (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal scar, new (Eye disorders) | 3 (4) | 5 (6) | 4 (5)
Solution induced corneal staining (Eye disorders) | 28 (28) | 35 (35) | 28 (28)
Poor contact lens fit (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Foreign body (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 5 (5) | 3 (3) | 5 (5)
Contact lens solution issue (Eye disorders) | 3 (3) | 2 (2) | 5 (5)
Conjunctivitis, any type (Eye disorders) | 5 (5) | 5 (5) | 5 (5)
Subconjunctival hemorrhage (Eye disorders) | 3 (3) | 2 (2) | 3 (3)
Retinal issue (Eye disorders) | 4 (4) | 2 (2) | 4 (4)
Optic nerve issue (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Trauma, ocular (Eye disorders) | 1 (1) | 0 (0) | 3 (3)
Binocular vision/accommodation issue (Eye disorders) | 5 (5) | 1 (1) | 5 (5)
Color vision defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Transient visual disturbance (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Unspecified contact lens issue (Eye disorders) | 1 (1) | 2 (2) | 3 (3)
Visual symptoms, no obvious cause (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Allergy, non-ocular (Immune system disorders) | 3 (3) | 1 (1) | 0 (0)
Trauma, non-ocular (General disorders) | 19 (21) | 12 (13) | 7 (9)
Headaches (General disorders) | 6 (7) | 3 (3) | 6 (7)
Concussion (General disorders) | 1 (1) | 1 (1) | 4 (4)
Systemic disease (General disorders) | 8 (8) | 9 (9) | 10 (12)
Mental health issues (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2)
Can't categorize (General disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form: University of Houston Informed Consent (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02255474/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT02255474/Prot_SAP_002.pdf
  • Informed Consent Form: Ohio State University Clinical Site (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02255474/ICF_003.pdf